CLINICAL TRIAL: NCT06754657
Title: Comparison of Continuous vs. Single-injection Interscalene Block on QoR-15 in Outpatient Rotator Cuff Surgery: A Randomized Study Assessing Non-inferiority and Superiority (CORA-Q15)
Brief Title: CORA-Q15: Continuous vs. Single-injection Interscalene Block on QoR-15 in Outpatient Rotator Cuff Surgery
Acronym: CORA-Q15
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 240829017
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-12

CONDITIONS: Arthropathy Shoulder; Pain, Acute; Anesthesia
Keywords: ambulatory surgery; rotator cuff repair; regional anesthesia
MeSH Terms: conditions — Acute Pain | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Randomized, blinded, two-group clinical trial with a two-stage analysis (non-inferiority followed by superiority, if applicable).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Due to the nature of the intervention, both patients and healthcare personnel involved in the intraoperative and postoperative care of the patients will be blinded to the intervention.
  The PCA button for administering rescue boluses will be stored inside an opaque bag, containing the pump and button, so it will not be available for initial use by the volunteers. The control group will have the infusion activated and the bolus button clamped, while the intervention group will have the infusion set to zero and the bolus button unclamped.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infusion (Active Comparator): Patients infusion rate will be set to 4 ml/h, with 5 ml boluses (30-minute lockout). The PCA button will be disabled for rescue bolus administration.
  Interventions: Procedure: Single injection
- Bolus (Experimental): Patients infusion rate will be set to 0 ml/h, with 5 ml boluses (30-minute lockout). The PCA button will be enabled for rescue bolus administration.
  Interventions: Procedure: Continuous perineural infusion

INTERVENTIONS:
Procedure: Continuous perineural infusion — infusion rate 4 ml/h, with 5 ml boluses (30-minute lockout). The PCA button disabled
  Arms: Bolus
Procedure: Single injection — infusion rate 0 ml/h, with 5 ml boluses (30-minute lockout). The PCA button will be enabled for rescue bolus administration
  Arms: Infusion

SUMMARY:
The purpose of the study will be to compare the efficacy of single-injection interscalene block versus continuous interscalene block on the quality of recovery in patients undergoing outpatient arthroscopic rotator cuff repair surgery.

The participants will:

* Be randomized to receive either a single-injection interscalene block or continuous infusion via an elastomeric pump.
* Be monitored via telephone by the research team to complete the QoR-15 survey, assess pain levels, the need for tramadol use, and any complications.
* Have follow-up by the Acute Pain Unit during the first 3 days.

DETAILED DESCRIPTION:
After obtaining approval from the institutional CEC-CCSS and prospective registration of the study at clinicaltrials.org, the investigators will recruit patients who meet the inclusion criteria and provide written consent.

Following surgery and placement of the interscalene block with a catheter, in the recovery unit, participants will be assigned to one of two groups according to a random number table, in a 1:1 ratio using block randomization (block sizes of 4, 6, and 8) through sealed envelopes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years, < 75 years) scheduled for elective outpatient arthroscopic rotator cuff repair surgery.
* Patients capable of managing a continuous outpatient regional analgesia system based on an interscalene block (eligibility criteria: able to understand verbal and written instructions, have home support, and live geographically close to the healthcare center).
* Willing and able to provide informed, written consent to participate in the study.

Exclusion Criteria:

* History of chronic opioid use (>3 months).
* Severe comorbidities (e.g., renal or hepatic failure, ASA classification of 3 or higher).
* Allergy to local anesthetics, dexamethasone, or the analgesic drugs used in the study.
* Patients with contraindications for peripheral nerve block.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Daily score on the "Quality of Recovery-15" (QoR-15) scale during the first 3 postoperative days. | Preoperative score and daily score during the first 3 postoperative days.
  The QoR-15 is a validated instrument in the literature that assesses the quality of recovery in patients after surgery. It is a multidimensional measurement tool that allows healthcare professionals to gain an overview of the patient's well-being during the postoperative period. The questionnaire consists of 15 items, covering 5 dimensions: Physical Comfort, Physical Independence, Emotional Support, Psychological Well-being, and Satisfaction with Recovery. The minimum score on the scale is 0 points, and the maximum score is 150 points. This range is obtained by summing the scores of the different categories evaluated in the QoR-15 scale, where a higher score indicates a better quality of postoperative recovery.

SECONDARY OUTCOMES:
Opioid consumption during the first 3 postoperative days | Daily consumption during the first 3 postoperative days.
  To assess rescue opioid consumption, expressed as morphine equivalents, during the first three postoperative days.
Daily Numeric Rating Score (NRS) during the first 3 postoperative days | Daily NRS during the first 3 postoperative days
  The NRS (Numeric Rating Scale) is commonly used to assess pain intensity. Its minimum score is 0, indicating no pain, and its maximum score is 10, indicating the worst pain imaginable. This scale is simple and allows patients to rate their pain using a number from 0 to 10. The objective is to assess the intensity of acute postoperative pain, expressed as NRS, during the first 3 postoperative days.
Rate of consultations/readmissions | During the first 3 postoperative days
  To assess the rate of consultations or readmissions due to pain or other complications in both groups.
Rate of rescue analgesic (bolus) during the first 3 postoperative days | During the first 3 postoperative days
  In the case that patients do not experience pain relief with the established management, as indicated by persistent NRS ≥ 4 after the administration of more than two rescue tramadol tablets, they will be instructed to call the contact phone number of the Ambulatory Pain Management Unit to receive guidance on how to implement a rescue bolus using the perineural catheter and the bolus option of the elastomeric pump. This event will be documented and recorded with the time of occurrence in a mobile application developed for this purpose.

CONTACTS AND LOCATIONS:
Locations (1):
- Red de Salud UC Christus, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chou LB, Wagner D, Witten DM, Martinez-Diaz GJ, Brook NS, Toussaint M, Carroll IR. Postoperative pain following foot and ankle surgery: a prospective study. Foot Ankle Int. 2008 Nov;29(11):1063-8. doi: 10.3113/FAI.2008.1063. PMID 19026197
- [Background] Joshi G, Gandhi K, Shah N, Gadsden J, Corman SL. Peripheral nerve blocks in the management of postoperative pain: challenges and opportunities. J Clin Anesth. 2016 Dec;35:524-529. doi: 10.1016/j.jclinane.2016.08.041. Epub 2016 Oct 20. PMID 27871587
- [Background] Neal JM, Gerancher JC, Hebl JR, Ilfeld BM, McCartney CJ, Franco CD, Hogan QH. Upper extremity regional anesthesia: essentials of our current understanding, 2008. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):134-70. doi: 10.1097/AAP.0b013e31819624eb. PMID 19282714
- [Background] Xu J, Chen XM, Ma CK, Wang XR. Peripheral nerve blocks for postoperative pain after major knee surgery. Cochrane Database Syst Rev. 2014;(12):CD010937. doi: 10.1002/14651858.CD010937.pub2. Epub 2014 Dec 11. PMID 25501884
- [Background] Ilfeld BM, Vandenborne K, Duncan PW, Sessler DI, Enneking FK, Shuster JJ, Theriaque DW, Chmielewski TL, Spadoni EH, Wright TW. Ambulatory continuous interscalene nerve blocks decrease the time to discharge readiness after total shoulder arthroplasty: a randomized, triple-masked, placebo-controlled study. Anesthesiology. 2006 Nov;105(5):999-1007. doi: 10.1097/00000542-200611000-00022. PMID 17065895
- [Background] Pehora C, Pearson AM, Kaushal A, Crawford MW, Johnston B. Dexamethasone as an adjuvant to peripheral nerve block. Cochrane Database Syst Rev. 2017 Nov 9;11(11):CD011770. doi: 10.1002/14651858.CD011770.pub2. PMID 29121400
- [Background] Lehmann N, Joshi GP, Dirkmann D, Weiss M, Gulur P, Peters J, Eikermann M. Development and longitudinal validation of the overall benefit of analgesia score: a simple multi-dimensional quality assessment instrument. Br J Anaesth. 2010 Oct;105(4):511-8. doi: 10.1093/bja/aeq186. Epub 2010 Aug 6. PMID 20693179
- [Background] Mascha EJ, Turan A. Joint hypothesis testing and gatekeeping procedures for studies with multiple endpoints. Anesth Analg. 2012 Jun;114(6):1304-17. doi: 10.1213/ANE.0b013e3182504435. Epub 2012 May 3. PMID 22556210
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Chazapis M, Walker EM, Rooms MA, Kamming D, Moonesinghe SR. Measuring quality of recovery-15 after day case surgery. Br J Anaesth. 2016 Feb;116(2):241-8. doi: 10.1093/bja/aev413. PMID 26787793
- [Background] Myles PS, Myles DB. An Updated Minimal Clinically Important Difference for the QoR-15 Scale. Anesthesiology. 2021 Nov 1;135(5):934-935. doi: 10.1097/ALN.0000000000003977. No abstract available. PMID 34543410
- [Background] Admiraal M, Smulders PSH, Rutten MVH, de Groot EK, Heine Y, Baumann HM, van der Vegt VHC, Halm JA, Hermanns H, Schepers T, Hollmann MW, Hermanides J, Ten Hoope W. The effectiveness of ambulatory continuous popliteal sciatic nerve blockade on patient-reported overall benefit of analgesia in patients undergoing foot or ankle surgery (CAREFREE trial); a randomized, open label, non-inferiority trial. J Clin Anesth. 2024 Aug;95:111451. doi: 10.1016/j.jclinane.2024.111451. Epub 2024 Apr 3. PMID 38574504
- [Background] Morales-Ariza V, Loaiza-Aldean Y, de Miguel M, Pena-Navarro M, Martinez-Silva O, Gonzalez-Tallada A, Manrique-Munoz S, de Nadal M. Validation and cross-cultural adaptation of the postoperative quality of recovery 15 (QoR-15) questionnaire for Spanish-speaking patients: A prospective cohort study. Am J Surg. 2023 Apr;225(4):740-747. doi: 10.1016/j.amjsurg.2022.11.009. Epub 2022 Nov 17. PMID 36414472
- [Background] Aliste J, Layera S, Bravo D, Aguilera G, Erpel H, Garcia A, Lizama M, Finlayson RJ, Tran D. Randomized comparison between perineural dexamethasone and combined perineural dexamethasone-dexmedetomidine for ultrasound-guided infraclavicular block. Reg Anesth Pain Med. 2022 Jun 21:rapm-2022-103760. doi: 10.1136/rapm-2022-103760. Online ahead of print. PMID 35728840